CLINICAL TRIAL: NCT02010593
Title: Phase 2a Safety Study of a Vaginal Matrix Ring Containing Dapivirine in a Postmenopausal Female Population
Brief Title: Safety and Pharmacokinetics of Dapivirine Vaginal Ring in Post-menopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MTN-024/IPM031; 5UM1AI068633-07 (NIH)
Record Dates: First submitted 2013-10-14; First posted 2013-12-13 (Estimated); Results first posted 2022-10-05 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Dapivirine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapivirine Vaginal Ring (Experimental): Safety study of a vaginal ring containing Dapivirine in a postmenopausal female population
  Interventions: Drug: Dapivirine Vaginal Ring
- Placebo (Placebo Comparator): The placebo VR is a flexible, platinum-catalyzed-cured matrix ring, identical to Dapivirine Ring-004, containing no active-drug
  Interventions: Drug: Placebo Vaginal Ring

INTERVENTIONS:
Drug: Dapivirine Vaginal Ring — Dapivirine, a non-nucleoside reverse-transcriptase inhibitor (NNRTI), is a substituted amino- pyrimidine (DAPY) derivative with potent antiviral activity against HIV-1. Dapivirine is chemically described as 4-[[4-[(2,4,6-trimethylphenyl)amino]-2- pyrimidinyl]amino]benzonitrile.6 The dapivirine matrix VR is a flexible ring containing 25 mg of drug substance dispersed in a platinum-catalyzed-cured silicone matrix. Dapivirine is known to be well-suited for delivery via VR
  Other Names: TMC-120
  Arms: Dapivirine Vaginal Ring
Drug: Placebo Vaginal Ring — The placebo VR is a flexible, platinum-catalyzed-cured silicone matrix ring, identical to dapivirine Ring-004, containing no active drug.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety of the dapivirine vaginal ring when inserts once every 4 weeks in postmenopausal women over 12 weeks of product use.

DETAILED DESCRIPTION:
Dapivirine, a non-nucleoside reverse-transcriptase inhibitor (NNRTI), is a substituted diamino- pyrimidine (DAPY) derivative with potent antiviral activity against HIV-1. Dapivirine is chemically described as 4-[[4-[(2,4,6-trimethylphenyl)amino]-2- pyrimidinyl]amino]benzonitrile.6 The dapivirine matrix VR is a flexible ring containing 25 mg of drug substance dispersed in a platinum-catalyzed-cured silicone matrix. Dapivirine is known to be well-suited for delivery via VR, as evidenced by favorable safety and pharmacokinetic data to date described below.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 through 65 years (inclusive) at Screening, verified per site SOPs
2. Per participant report, postmenopausal at Screening, defined as amenorrhoeic for the past 12 months (minimum) or at least 6 months status post-bilateral oophorectomy
3. Follicle-stimulating hormone (FSH) level at 40 mIU/ml or higher at Screening
4. Able and willing to provide written informed consent to be screened for and enrolled in MTN-024/IPM 031
5. Able to communicate in spoken and written English
6. Able and willing to comply with all study procedural requirements
7. Willing to only use study provided and/or approved vaginal products throughout the duration of study participation.
8. Willing to abstain from inserting study approved lubricant into the vagina for 72 hours prior to each visit
9. Willing to abstain from vaginal intercourse for 72 hours prior to each visit
10. In general good health as determined by the Investigator of Record (IoR)/designee at Screening and Enrollment
11. Able and willing to provide adequate locator information, as defined in site SOPs
12. HIV-uninfected based on testing performed at Screening (per protocol algorithm in Appendix II)
13. Per participant report at Screening and Enrollment, agrees to use male latex condoms for sexual intercourse
14. Per participant report at Screening and Enrollment, states a willingness to refrain from inserting any non-study vaginal products or objects into the vagina including, but not limited to spermicides, female condoms, diaphragms, topical or systemic hormone replacement therapy, including vaginal estrogens, and/or hormonal contraceptives, vaginal medications, menstrual cups, cervical caps (or any other vaginal barrier method), vaginal douches, lubricants and moisturizers, sex toys (vibrators, dildos, etc.), for the duration of the study participation.

    Note: Use of study approved lubricant is permitted.
15. At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products, or vaccines for the duration of study participation

    Participants in the biopsy subset must also meet the following criteria at Screening to be eligible for inclusion:
16. Willing to abstain from inserting anything into the vagina for 72 hours following the collection of biopsies, including abstaining from vaginal intercourse
17. Anatomy sufficient for the collection of cervical biopsies

Exclusion Criteria:

1. Per participant report at screening:

   1. Plans to relocate away from the study site during study participation
   2. Plans to travel away from the study site for more than 4 consecutive weeks during study participation
2. Pregnant at screening Note: A documented negative pregnancy test performed by study staff is required for inclusion; however a self-reported pregnancy is adequate for exclusion from the study.
3. Diagnosed with urinary tract infection (UTI) at Screening or Enrollment Note: Otherwise eligible participants diagnosed with UTI during screening are offered treatment and may be enrolled after completing treatment and all symptoms have resolved.

   If treatment is completed and symptoms have resolved within 45 days of obtaining informed consent for screening, the participant may be enrolled.
4. Diagnosed with pelvic inflammatory disease, an STI or reproductive tract infection (RTI) requiring treatment per current Centers for Disease Control and Prevention (CDC) guidelines at Screening or Enrollment Note: Otherwise eligible participants diagnosed during screening with pelvic inflammatory disease or STI/RTI requiring treatment per CDC guidelines - other than asymptomatic bacterial vaginosis (BV) and asymptomatic candidiasis - are offered treatment and may be enrolled after completing treatment and all symptoms have resolved. If treatment is completed and symptoms have resolved within 45 days of obtaining informed consent for screening, the participant may be enrolled. Genital warts requiring treatment also must be treated prior to Enrollment. Genital warts requiring therapy are defined as those that cause undue burden or discomfort to the participant, including bulky size, unacceptable appearance, or physical discomfort.
5. Has a clinically apparent Grade 2 or higher pelvic exam finding (observed by study staff) at Screening or Enrollment, as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009), Addendum 1-Female Genital Grading Table for Use in Microbicide Studies Note: Cervical bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the Investigator of Record (IoR)/designee is considered expected non-menstrual bleeding and is not exclusionary.

   Note: Otherwise eligible participants with exclusionary pelvic exam findings may be enrolled/randomized after the findings have improved to a non-exclusionary severity grading or resolved. If improvement to a non-exclusionary grade or resolution is documented within 45 days of providing informed consent for screening, the participant may be enrolled.
6. Participant report and/or clinical evidence of any of the following:

   1. Known adverse reaction to any of the study products (ever)
   2. Known adverse reaction to latex (ever)
   3. Chronic and/or recurrent vaginal candidiasis
   4. Topical or systemic hormone replacement therapy and/or hormonal contraception within the 6 months prior to Enrollment
   5. Non-therapeutic injection drug use in the 12 months prior to Enrollment
   6. Post-exposure prophylaxis (PEP) for HIV exposure within the 6 months prior to Enrollment
   7. Pre-exposure prophylaxis (PrEP) for HIV prevention within the 6 months prior to Enrollment
   8. Last pregnancy outcome 6 months or less prior to Enrollment
   9. Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage, piercing) 90 days or less prior to Enrollment
   10. Currently breastfeeding
   11. At Screening, severe pelvic relaxation such that either the vaginal walls or the uterine cervix descend beyond the vaginal introitus with Valsalva maneuver
   12. Participation in any other research study involving drugs, medical devices, vaginal products, or vaccines, in the 45 days prior to Enrollment
7. As determined by the IoR/designee, any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease
8. Has any of the following laboratory abnormalities at Screening Visit:

   1. Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher*
   2. Creatinine Grade 2 or higher*
   3. Hemoglobin Grade 2 or higher*
   4. Platelet count Grade 1 or higher*
   5. Pap result Grade 2 or higher** Note: Otherwise eligible participants with an exclusionary test may be re-tested during the screening process.

   Note: Women with a documented normal result within the 12 months prior to Enrollment need not have a Pap smear during the screening period. Women with a Grade 1 abnormal Pap smear can be enrolled upon completion of the initial phase of evaluation if no current treatment is indicated (based on local standard of care for management of abnormal cervical cytology). Need for a repeat Pap within 6 months does not preclude Enrollment prior to that result becoming available. If the participant has had a hysterectomy for reasons not related to cervical dysplasia, a Pap smear need not be performed.
9. Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate the interpretation of study outcome data, or otherwise interfere with achieving the study objectives *Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 1.0, December, 2004 (Clarification dated August 2009) **Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the Division of AIDS (DAIDS) Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Alabama CRS, 84519th Street South, BBRB 203A, Birmingham, Alabama
  - Case CRS, Case Western Reserve University, 2061 Cornell Road, Room 303, Cleveland, Ohio
  - Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shapley-Quinn MK, Laborde N, Luecke E, Hoesley C, Salata RA, Johnson S, Nel A, Soto-Torres L, Chen BA, van der Straten A. Acceptability of the Dapivirine Vaginal Ring in Postmenopausal US Women. AIDS Patient Care STDS. 2022 Mar;36(3):97-105. doi: 10.1089/apc.2022.0002. PMID 35289688
- [Derived] Chen BA, Zhang J, Gundacker HM, Hendrix CW, Hoesley CJ, Salata RA, Dezzutti CS, van der Straten A, Hall WB, Jacobson CE, Johnson S, McGowan I, Nel AM, Soto-Torres L, Marzinke MA; MTN-024/IPM 031 Protocol Team for the Microbicide Trials Network. Phase 2a Safety, Pharmacokinetics, and Acceptability of Dapivirine Vaginal Rings in US Postmenopausal Women. Clin Infect Dis. 2019 Mar 19;68(7):1144-1151. doi: 10.1093/cid/ciy654. PMID 30289485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial staff pre-screened potential participants at either on-site or off-site locations. During these interactions, staff explained the trial to participants, ascertained elements of presumptive eligibility. Process info was recorded and stored in the absence of written IC from participants, provided the info was collected in such a manner that it could not be linked to participant identifiers.
  Participants were recruited at 3 medical centres between 23 Dec 2013 and 31 Dec 2014.
Pre-assignment Details: Two hundred participants provided written informed consent and were subsequently screened. Of these, 96 participants met recruitment criteria and were randomized.
Period: Overall Study
Arm/Group | Dapivirine Vaginal Ring | Placebo
Started | 72 | 24
Completed | 70 | 22
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Unable to adhere to visit schedule | 0 | 2

BASELINE CHARACTERISTICS:
Population: Sexually active, HIV-uninfected, postmenopausal women who was able to give written informed consent
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapivirine Vaginal Ring | Placebo | Total
Number analyzed (Participants) | 72 | 24 | 96
Age, Customized [Mean (Standard Deviation); unit: years]
  Age 45 - 65 (inclusive) | 57.2 (4.3) | 55.3 (3.0) | 56.8 (41.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 24 | 96
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 71 | 24 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 8 | 30
  White | 48 | 15 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 24 | 96
Main cause of menopause [Count of Participants; unit: Participants]
  Spontaneous | 60 | 18 | 78
  Surgical | 3 | 3 | 6
  Unknown | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety of Dapivirine (25 mg) Administered in a Silicone Elastomer Vaginal Matrix Ring in HIV-uninfected Postmenopausal Women, When Inserted Once Every 4 Weeks During 12 Weeks of Study Product Use
Description: Evidence of Grade 2 or higher genital, genitourinary and reproductive system AEs as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 (Clarification dated August 2009), Addendum 1, (Female Genital Grading Table for Use in Microbicide Studies) judged to be related to study product.
  Evidence of Grade 3 or higher AEs as defined by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Dec 2004 (Clarification dated August 2009).
  DAIDS severity grades are defined as follows:
  * Grade 1 = mild
  * Grade 2 = moderate
  * Grade 3 = severe
  * Grade 4 = potentially life-threatening
  * Grade 5 = death
Time Frame: over 12-week period of use
Population: Intent-to-Treat: All participants randomized in the trial were included in the primary analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo
Number analyzed (Participants) | 72 | 24
Participants
  DAIDS Grade 2 or higher | 6 | 3
  DAIDS grade 3 | 4 | 0

2. Secondary Outcome: The Percentage of Participants Who Find the Study Vaginal Ring to be as Acceptable
Description: To evaluate the acceptability, the percentage of participants who at their 12-Week Final Clinic Visit report via acceptability questionnaire that they prefer the ring at least as much as other HIV prevention methods.
Time Frame: at 12-week visit
Population: Participants who have answered to preference question at the week 12 visit
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo
Number analyzed (Participants) | 69 | 22
Participants | 61 | 20

3. Secondary Outcome: Percentage of Women Who Were Adherent to Daily Study Product Use Based on Self-report Over the 12-week Study Product Use Period
Description: Adherence will be measured by the percentage of women who keep the VR inserted at all times in the vagina over the course of 12 weeks.
  A participant was considered adherent in one month (4 weeks) by self-reported data, only if the ring was never out during that month and the participant was not on product hold and did not terminate the clinical trial within that month.
Time Frame: 12-week period of use
Population: Adherent Participant: based on self report, IP was never out during one month (4 week)
Measure: Count of Participants; unit: Participants
Arm/Group | Dapivirine Vaginal Ring | Placebo
Number analyzed (Participants) | 72 | 24
Participants
  Week 0 - 4 | 58 | 22
  Week 4 - 8 | 67 | 22
  Week 8 - 12 | 65 | 21

4. Secondary Outcome: Pharmacokinetics - The Intent is to Determine if the Plasma Dapivirine Concentrations Are Different in Postmenopausal Women Than in Pre-menopausal Adult Women After Placement of Dapivirine Vaginal Rings.
Description: The PK endpoint is a description of the end of period (28 day post ring insertion) plasma dapivirine concentrations at week 4, 8, and 12 which will be compared to the same results in a recently studied population of premenopausal adult women (MTN-013).
Time Frame: a 12 week product use period
Population: The PK analysis population included all participants who were randomised to the active IP arm with a detectable concentration in plasma at any time during follow-up. One participant was not included in the PK analysis since she was terminated from the trial early (after Week 4) due to non-compliance. Four of these participants (71) had undetectable dapivirine concentrations in plasma samples in one or more visits:
  Week 4: 2 x participants Week 8: 1 x participant Week 12: 2 x participants
Measure: Mean (Standard Deviation); unit: picograms/mililiter
Arm/Group | Dapivirine Vaginal Ring
Number analyzed (Participants) | 71
picograms/mililiter
  Week 4: number analyzed (Participants) | 69
  Week 4 | 273.5 (98.2)
  Week 8: number analyzed (Participants) | 70
  Week 8 | 289.0 (123.8)
  Week 12: number analyzed (Participants) | 69
  Week 12 | 298.2 (143.2)

5. Secondary Outcome: Pharmacokinetics - The Intent is to Determine if the Vaginal Fluid Dapivirine Concentrations Are Different in Postmenopausal Women Than in Pre-menopausal Adult Women After Placement of Dapivirine Vaginal Rings.
Description: The PK endpoint is a description of the end of period (28 day post ring insertion) vaginal fluid dapivirine concentrations at week 4, 8, and 12 which will be compared to the same results in a recently studied population of premenopausal adult women (MTN-013).
Time Frame: a 12 week product use period
Population: PK analysis population included all participants who were randomised to active IP arm with a detectable concentration in vaginal fluid at any time during f/u.
  Results from 36 participants enrolled in dapivirine arm were available for analysis in vaginal fluid sample subset. For 35 participants, detectable dapivirine concentrations were measured in vaginal fluid at any time during f/u. 5 x participants had undetectable dapivirine concentrations in vaginal fluid samples in one or more visits.
Measure: Mean (Standard Deviation); unit: nanogram/miligram
Arm/Group | Dapivirine Vaginal Ring
Number analyzed (Participants) | 36
nanogram/miligram
  Week 4: number analyzed (Participants) | 33
  Week 4 | 64.3 (65.9)
  Week 8: number analyzed (Participants) | 34
  Week 8 | 78.5 (92.2)
  Week 12: number analyzed (Participants) | 33
  Week 12 | 72.1 (80)

ADVERSE EVENTS:
Time Frame: IP 12 weeks + 1 week follow-up
Description: All AEs (including deaths and SAE) reported by or observed in enrolled trial participants regardless of severity and presumed relationship to IP was reported in source documents.
Arm/Group | Dapivirine Vaginal Ring | Placebo
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/24
Other Adverse Events (participants affected / at risk) | 46/72 | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapivirine Vaginal Ring (N=72) | Placebo (N=24)
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Vaginal Ring (N=72) | Placebo (N=24)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3)
Vulvovaginitis (Infections and infestations) | 2 (2) | 2 (2)
Blood pressure increased (Investigations) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 8 (8) | 3 (3)
Vaginal erosion (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Vaginal odour (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulvovaginal erythema (Reproductive system and breast disorders) | 2 (3) | 3 (3)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The AEs reported were not unexpected in post-menopausal women. Due to the lack of a non-interventional arm or observational period, however, an objective evaluation of possible genital tract AEs associated with vaginal ring (VR) use could not be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes